CLINICAL TRIAL: NCT05356806
Title: Incidence of Peri-implant Mucositis in Patients With Treated Periodontitis: a Prospective Study.
Brief Title: Incidence of Peri-implant Mucositis in Patients With Treated Periodontitis
Acronym: PiM_Inc
Status: Recruiting | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Sociedad Española de Periodoncia (SEPA) (Unknown); Dentaid SL (Industry)
Responsible Party: Sponsor
Other Study IDs: 52-240521
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Peri-implant Mucositis
Keywords: peri-implant mucositis; incidence; biofilm; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples containing bacterial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One: Patients with treated periodontitis who have had dental implants placed at the Periodontics Specialist Clinic of the UCM School of Dentistry, and are going to be rehabilitated.
  Interventions: Other: Supportive periodontal and periimplant care

INTERVENTIONS:
Other: Supportive periodontal and periimplant care — Periodontal and peri-implant maintenance therapy will be carried out at baseline, 3 and 6-month visit. This session will include the removal of biofilm and calculus on teeth and implants (except those that have just been restored) with an ultrasonic device using a plastic tip ( for implants. and a conventional metal tip ( for teeth. At the end, polishing will be done with a rubber cup
  Subsequently, patients will be explained that they must continue with their usual oral hygiene technique on their teeth, using the same type of brush (which can be electric or manual), interproximal devices, toothpaste or mouthwash used to date. Finally, they will receive specific instructions for the supragingival biofilm control in the area of the new restoration and will be given interdental brushes that suit to the space

SUMMARY:
the objective of this study is to determine the incidence of peri-implant mucositis in patients with treated periodontitis and enrolled in periodontal maintenance and to evaluate the associated risk indicators. An analytical prospective observational study will be carried out, with an initial follow-up of 12 months.

DETAILED DESCRIPTION:
Introduction: Peri-implant mucositis (PM) is an inflammatory disease induced by the accumulation of bacteria (biofilm) around dental implants, which can be modulated by individual characteristics of the patient, as well as by numerous factors related to a greater accumulation of biofilm in peri-implant tissues. Without correct regular maintenance, this entity can progress to peri-implantitis, a disease in which there is loss of bone supporting the implant. However, the strength of the association of the factors with the appearance of PM remains weak and incidence studies are limited due to their design and methodological inconsistencies. Therefore, the objective of this study is to determine the incidence of PM in patients with treated periodontitis and enrolled in periodontal maintenance and to evaluate the associated risk indicators.

Material and method: An analytical prospective observational study will be carried out, with an initial follow-up of 12 months. Patients with treated periodontitis and enrolled in periodontal maintenance will be selected, consecutively. They need to have implants placed in the Periodontics Specialist Clinic and are going to be rehabilitated at the UCM School of Dentistry. Peri-implant and periodontal clinical records, radiographic records, demographic variables, patient-based variables, and submucosal microbiological samples will be taken on the day of crown placement and after 6 and 12 months. The calculation of the sample size estimates the need to recruit 227 patients. The results will be analyzed using regression models.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, able to comply with the protocol and comply with the established visits.
* Patients with treated periodontitis and enrolled in periodontal maintenance (last maintenance therapy received between 4 and 6 months maximum before inclusion in the study) (Chapple et al., 2018, Sanz et al., 2020).
* Patients with osseointegrated dental implants waiting for their prosthodontic rehabilitation (fixed prosthesis [individual, partial or complete], hybrid or overdenture).
* Physical or mental conditions that make it possible to perform appropiate oral hygiene

Exclusion Criteria:

* Patients with untreated periodontitis.
* Totally edentulous patients.
* Patients with peri-implant diseases.
* Pregnant or in lactating-period patients.
* Patients undergoing treatment with medication that affects the periodontal/peri-implant status or the immune system (phenytoin, calcium antagonists, corticosteroids or anti-inflammatories).
* Patients who have taken antibiotics in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treated periodontitis who have had dental implants placed at the Periodontics Specialist Clinic of the UCM School of Dentistry, and are going to be rehabilitated in the same center
Sampling Method: Non-Probability Sample
Enrollment: 277 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of peri-implant mucositis | 12 months
  The risk of developing PM (patient with at least one implant who has bleeding on probing, with or without suppuration and without progressive radiographic bone loss) during a follow-up period of 12 months.

SECONDARY OUTCOMES:
Affiliation data | Baseline
  Age, Sex
previous medical history | Baseline
  systemic diseases, medication, allergies
smoking habit | Baseline
  ex-smoker/smoker/non-smoker
Other general data | Baseline
  sports habit, educational level, alcohol and coffee consumption, type of diet.
Previous dental history | Baseline
  history of periodontitis, periodontal treatment received (date of maintenance therapy, basic or surgical treatment), as well as the presence of previous peri-implant diseases will be recorded. Toothbrushing device used by the patient (manual or electric toothbrush) will also be recorded.
Characteristics of the teeth that have been replaced by implants | Baseline
  Options:single tooth in the anterior region, single tooth in the posterior region, tooth with distal extension, interdental space, edentulous upper jaw, edentulous lower jaw
Surgical procedure | Baseline
  bone regeneration procedures (prior, simultaneous, immediate implant), alveolar preservation, use of platelet derivatives, use of bone graft (autologous, xenogenic, mixed), use of membranes, sinus lift or soft tissue augmentation.
Implant characteristics | Baseline
  location (maxillary, mandibular, both), implant system (brand, implant position relative to bone and soft tissue, platform change, configuration, implant material), surface topography (roughness index), diameter and length (measured in millimeters),
Characteristics of the restorations | Baseline
  existence or not of an intermediate abutment and its characteristics, retention of the crown (cemented, screw-retained, cement-retained or other), type of prosthetic restoration (fixed prosthesis [individual, partial or complete], hybrid or overdenture ), crown material (metal-porcelain, ceramic, zirconium or resin), crown design method (CAD-CAM/casting) and impression-taking method (intraoral scanner, registration with silicone measurements) and if there are clinical signs of bruxism
Mucosal thickness (GM) | Baseline
  it will be measured with a K45 file (Stainless Steal K-File, Dentsply Maillefer, Ballaigues, Switzerland) and PCP15 periodontal probe calibrated in millimeters (HuFriedy® , Chicago, IL, USA), 1 mm from mucosal margin and at the buccal and lingual center of each implant.
Mucosal height | Baseline
  (once the abutment/healing screw has been removed, before placing the restoration): distance from the margin of the peri-implant mucosa to the implant head. It will be measured with a PCP15 periodontal probe calibrated in millimeters (HuFriedy®, Chicago, IL, USA), in 6 locations for each implant.
Modified plaque index (mPI) | Baseline
  Score 0: no plaque detected; score 1: plaque is only recognized by passing a probe over the smooth marginal surface of the implant; score 2: the plaque is visible; score 3: abundance of soft plaque.
Modified plaque index (mPI) | 6 months
  Score 0: no plaque detected; score 1: plaque is only recognized by passing a probe over the smooth marginal surface of the implant; score 2: the plaque is visible; score 3: abundance of soft plaque.
Modified plaque index (mPI) | 12 months
  Score 0: no plaque detected; score 1: plaque is only recognized by passing a probe over the smooth marginal surface of the implant; score 2: the plaque is visible; score 3: abundance of soft plaque.
Modified sulcus bleeding Index (mBI) | Baseline
  Score 0: no bleeding when passing a periodontal probe along the mucosal margin adjacent to the implant; score 1: visible isolated bleeding point; score 2: the bleed forms a confluent red line in the margin; score 3: profuse bleeding.
Modified sulcus bleeding Index (mBI) | 6 months
  Score 0: no bleeding when passing a periodontal probe along the mucosal margin adjacent to the implant; score 1: visible isolated bleeding point; score 2: the bleed forms a confluent red line in the margin; score 3: profuse bleeding.
Modified sulcus bleeding Index (mBI) | 12 months
  Score 0: no bleeding when passing a periodontal probe along the mucosal margin adjacent to the implant; score 1: visible isolated bleeding point; score 2: the bleed forms a confluent red line in the margin; score 3: profuse bleeding.
Bleeding on probing (BOP) | Baseline
  assessed dichotomously within 15 seconds of probing. Bleeding must be clear (a spot bleed will not be considered positive).
Bleeding on probing (BOP) | 6 months
  assessed dichotomously within 15 seconds of probing. Bleeding must be clear (a spot bleed will not be considered positive).
Bleeding on probing (BOP) | 12 months
  assessed dichotomously within 15 seconds of probing. Bleeding must be clear (a spot bleed will not be considered positive).
Suppuration on probing (Sup): | Baseline
  evaluated dichotomously after probing.
Suppuration on probing (Sup): | 6 months
  evaluated dichotomously after probing.
Suppuration on probing (Sup): | 12 months
  evaluated dichotomously after probing.
Probing depth (PS) | Baseline
  defined as the distance in mm between the depth of the pocket and the margin of the peri-implant tissue.
Probing depth (PS) | 6 months
  defined as the distance in mm between the depth of the pocket and the margin of the peri-implant tissue.
Probing depth (PS) | 12 months
  defined as the distance in mm between the depth of the pocket and the margin of the peri-implant tissue.
Crown length (CL): | Baseline
  defined as the distance, in mm, between the incisal/occlusal part of the crown and the margin of the peri-implant tissue.
Crown length (CL): | 6 months
  defined as the distance, in mm, between the incisal/occlusal part of the crown and the margin of the peri-implant tissue.
Crown length (CL): | 12 months
  defined as the distance, in mm, between the incisal/occlusal part of the crown and the margin of the peri-implant tissue.
Width of the mucosa: | Baseline
  distance from the mucosal margin to the mucogingival line at the buccal and lingual center. It will be measured with a PCP15 periodontal probe calibrated in millimeters (HuFriedy®, Chicago, IL, USA).
Width of the mucosa: | 6 months
  distance from the mucosal margin to the mucogingival line at the buccal and lingual center. It will be measured with a PCP15 periodontal probe calibrated in millimeters (HuFriedy®, Chicago, IL, USA).
Width of the mucosa: | 12 months
  distance from the mucosal margin to the mucogingival line at the buccal and lingual center. It will be measured with a PCP15 periodontal probe calibrated in millimeters (HuFriedy®, Chicago, IL, USA).
full-mouth periodontal clinical parameters | Baseline
  will be recorded at 6 locations per tooth and implant with a PCP15 periodontal probe (HuFriedy®, Chicago, IL, USA). These include PS, recession (REC), BOP, clinical attachment level (CAL), plaque index (PI), Sup.
full-mouth periodontal clinical parameters | 6 months
  will be recorded at 6 locations per tooth and implant with a PCP15 periodontal probe (HuFriedy®, Chicago, IL, USA). These include PS, recession (REC), BOP, clinical attachment level (CAL), plaque index (PI), Sup.
full-mouth periodontal clinical parameters | 12 months
  will be recorded at 6 locations per tooth and implant with a PCP15 periodontal probe (HuFriedy®, Chicago, IL, USA). These include PS, recession (REC), BOP, clinical attachment level (CAL), plaque index (PI), Sup.
Radiographic bone level | Baseline
  defined as the distance between the implant shoulder and the first visible contact between the implant surface and the most apical position of the bone in mesial and distal. For transmucosal implants, the length of the intermediate abutment will not be taken into account. Implant distances (length and diameter) will be used for fit and distortion. In visit 1, a perpendicular line to the major axis of the implant will be drawn, coinciding with the position of the bone level, this reference will be the guide to assess possible discrepancies in the following visits.
Radiographic bone level | 6 months
  defined as the distance between the implant shoulder and the first visible contact between the implant surface and the most apical position of the bone in mesial and distal. For transmucosal implants, the length of the intermediate abutment will not be taken into account. Implant distances (length and diameter) will be used for fit and distortion. In visit 1, a perpendicular line to the major axis of the implant will be drawn, coinciding with the position of the bone level, this reference will be the guide to assess possible discrepancies in the following visits.
Radiographic bone level | 12 months
  defined as the distance between the implant shoulder and the first visible contact between the implant surface and the most apical position of the bone in mesial and distal. For transmucosal implants, the length of the intermediate abutment will not be taken into account. Implant distances (length and diameter) will be used for fit and distortion. In visit 1, a perpendicular line to the major axis of the implant will be drawn, coinciding with the position of the bone level, this reference will be the guide to assess possible discrepancies in the following visits.
Implant-Abutment Gap | Baseline
  Presence of space between implant and abutment and excess cement (surrounding excess cement will be explored).
Implant-Abutment Gap | 6 months
  Presence of space between implant and abutment and excess cement (surrounding excess cement will be explored).
Implant-Abutment Gap | 12 months
  Presence of space between implant and abutment and excess cement (surrounding excess cement will be explored).
Emergence angle and profile (concave/straight or convex) of restorations | Baseline
  The angle of the restoration will be measured mesial and distal according to the criteria established by Yotnuengnit et al. (Yotnuengnit et al., 2008). The emergence of the angle will be calculated between the length of the major axis of the implant and the tangent line to the restoration, then a tangential line is made from the restoration to the platform, the intersection angle is measured as an emergency angle. These measurements will be repeated twice for each mesial and distal surface. Each emergence profile will be categorized as concave, straight, or convex. For implants placed at bone level, the transmucosal abutment will be considered as a part of the restoration. According to this criterion, restorations with at least a 30º angle will be considered "over-contoured" (Kohal et al., 2003). Concave, convex and straight profile categories will awarded according to this emergency.
Emergence angle and profile (concave/straight or convex) of restorations | 6 months
  The angle of the restoration will be measured mesial and distal according to the criteria established by Yotnuengnit et al. (Yotnuengnit et al., 2008). The emergence of the angle will be calculated between the length of the major axis of the implant and the tangent line to the restoration, then a tangential line is made from the restoration to the platform, the intersection angle is measured as an emergency angle. These measurements will be repeated twice for each mesial and distal surface. Each emergence profile will be categorized as concave, straight, or convex. For implants placed at bone level, the transmucosal abutment will be considered as a part of the restoration. According to this criterion, restorations with at least a 30º angle will be considered "over-contoured" (Kohal et al., 2003). Concave, convex and straight profile categories will awarded according to this emergency.
Emergence angle and profile (concave/straight or convex) of restorations | 12 months
  The angle of the restoration will be measured mesial and distal according to the criteria established by Yotnuengnit et al. (Yotnuengnit et al., 2008). The emergence of the angle will be calculated between the length of the major axis of the implant and the tangent line to the restoration, then a tangential line is made from the restoration to the platform, the intersection angle is measured as an emergency angle. These measurements will be repeated twice for each mesial and distal surface. Each emergence profile will be categorized as concave, straight, or convex. For implants placed at bone level, the transmucosal abutment will be considered as a part of the restoration. According to this criterion, restorations with at least a 30º angle will be considered "over-contoured" (Kohal et al., 2003). Concave, convex and straight profile categories will awarded according to this emergency.
Patient reported outcomes | Baseline
  It will be recorded if the patient reports the appearance of pain in peri-implant tissues (no pain/slight pain/moderate pain/severe pain), need of analgesia (yes/no), inflammation (no inflammation/inflammation not visually perceived/evident inflammation) , bleeding (no bleeding/incipient bleeding when brushing/profuse bleeding when brushing), discomfort during brushing (no pain/slight pain/moderate pain/severe pain), collaboration (number of tooth brushings per day), oral hygiene habits (use of interproximal devices in the implants under study).
  In addition, type of toothbrush (manual/electric/sonic) and its frequency, use of dental floss (yes/no), use of interproximal brushes (yes/no) and use of mouthrinse (yes/no; frequency, type of mouthwash).
Patient reported outcomes | 6 months
  It will be recorded if the patient reports the appearance of pain in peri-implant tissues (no pain/slight pain/moderate pain/severe pain), need of analgesia (yes/no), inflammation (no inflammation/inflammation not visually perceived/evident inflammation) , bleeding (no bleeding/incipient bleeding when brushing/profuse bleeding when brushing), discomfort during brushing (no pain/slight pain/moderate pain/severe pain), collaboration (number of tooth brushings per day), oral hygiene habits (use of interproximal devices in the implants under study).
  In addition, type of toothbrush (manual/electric/sonic) and its frequency, use of dental floss (yes/no), use of interproximal brushes (yes/no) and use of mouthrinse (yes/no; frequency, type of mouthwash).
Patient reported outcomes | 12 months
  It will be recorded if the patient reports the appearance of pain in peri-implant tissues (no pain/slight pain/moderate pain/severe pain), need of analgesia (yes/no), inflammation (no inflammation/inflammation not visually perceived/evident inflammation) , bleeding (no bleeding/incipient bleeding when brushing/profuse bleeding when brushing), discomfort during brushing (no pain/slight pain/moderate pain/severe pain), collaboration (number of tooth brushings per day), oral hygiene habits (use of interproximal devices in the implants under study).
  In addition, type of toothbrush (manual/electric/sonic) and its frequency, use of dental floss (yes/no), use of interproximal brushes (yes/no) and use of mouthrinse (yes/no; frequency, type of mouthwash).
Microbiological samples | Baseline
  2 most accessible and/or inflamed locations will be selected. After careful removal of supramucosal biofilm deposits, if any, the areas of interest will be isolated using cotton rolls and air drying. Two sterile paper points (#30, Maillefer, Ballaigues, Switzerland) will be consecutively inserted into the peri-implant sulcus for 30 seconds. Paper points taken from each implant will be placed in a sterile and empty vial and will be sent within a maximum period of 24 hours to the research laboratory of the UCM School of Dentistry for subsequent freezing and processing (Pulcini et al., 2019 ). Analysis of the microbiome using massive sequencing techniques
Microbiological samples | 6 months
  2 most accessible and/or inflamed locations will be selected. After careful removal of supramucosal biofilm deposits, if any, the areas of interest will be isolated using cotton rolls and air drying. Two sterile paper points (#30, Maillefer, Ballaigues, Switzerland) will be consecutively inserted into the peri-implant sulcus for 30 seconds. Paper points taken from each implant will be placed in a sterile and empty vial and will be sent within a maximum period of 24 hours to the research laboratory of the UCM School of Dentistry for subsequent freezing and processing (Pulcini et al., 2019 ). Analysis of the microbiome using massive sequencing techniques
Microbiological samples | 12 months
  2 most accessible and/or inflamed locations will be selected. After careful removal of supramucosal biofilm deposits, if any, the areas of interest will be isolated using cotton rolls and air drying. Two sterile paper points (#30, Maillefer, Ballaigues, Switzerland) will be consecutively inserted into the peri-implant sulcus for 30 seconds. Paper points taken from each implant will be placed in a sterile and empty vial and will be sent within a maximum period of 24 hours to the research laboratory of the UCM School of Dentistry for subsequent freezing and processing (Pulcini et al., 2019 ). Analysis of the microbiome using massive sequencing techniques

CONTACTS AND LOCATIONS:
Overall Officials: Elena Figuero, Prof., Principal Investigator — Etiology and Therapy of Periodontal and Periimplant Research Group (ETEP). Faculty of Dentistry. University Complutense of Madrid (UCM)
Locations (1):
- Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No